CLINICAL TRIAL: NCT02862353
Title: Thrombocytopenia Drug Immune Validation of New Biological Test Diagnostic
Acronym: TITIM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1608040; 2016-A00858-43 (Other: ANSM)
Record Dates: First submitted 2016-07-29; First posted 2016-08-11 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Thrombocytopenia
Keywords: Validation new test
MeSH Terms: conditions — Thrombocytopenia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 dry tube of 5 ml for TITIM test
  1 dry tube of 7 ml for MAIPA test
  1 dry tube of 5 ml for serum bank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with thrombocytopenia drug
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — 15 ml of blood

SUMMARY:
The drug immune thrombocytopenia (TIM) are the most common drug cytopenias. They result from a peripheral destruction of platelets in the presence of the drug only. They usually involve immunoglobulin G (IgG) directed against either the drug molecule bound to a carrier protein or, by autoimmunity, against a hidden epitope newly exposed as a result of treatment. The most common drugs involved are quinine, some antibiotics, nonsteroidal anti-inflammatory drugs or anticonvulsants but the list is not exhaustive.

in the case of new-onset thrombocytopenia and after eliminating other possible causes, a TIM is suspected but the offending drug is difficult to identify in generally poly-medicated patients.

Several drugs may be suspected and the clinician uses biology for rapid assistance to the "de-prescription" and reduces unnecessary therapeutic substitutions in an always difficult clinical situation.

The Immunology Laboratory of the University Hospital of Saint-Etienne has developed a biological test of thrombocytopenia induction in the presence of the drug and the patient's serum that is to say its antibodies and complement fractions with cytometry reading flow. This Induction Test in vitro TIM (TITIM) is simple, fast, inexpensive, easy to transfer in hospital laboratories. But this test must be validated on well-documented clinical cases.

The purpose of this pilot project is to validate the technical and assess the clinical specificity of the test TITIM for hard imputability drugs validated by a committee of experts combining a posteriori of clinical and biological criteria of routine.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients with suspicion of thrombocytopenia drug
* consent signed

Exclusion Criteria:

* Thrombocytopenia plants such as secondary to the following molecules: antineoplastic (except oxaliplatin which gives TIM), immunosuppressants.
* Induced thrombocytopenia heparin and IIb / IIIa glycoproteins (abciximab, tirofiban, epifibatide).
* Presence of anti platelet antibodies allogeneic or autoimmune which are part of the MAIPA test.
* Patient exposed to at least one suspect molecule does not exist in water-soluble form or drug to which the metabolite is suspected
* Patients transfused (plasma, platelets) for less than a month
* Patients with an other bloodline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with thrombocytopenia drug
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
TITIM test positivity | at baseline
  TITIM test is considered positive when there is a decrease in platelet counts at least 10%.

CONTACTS AND LOCATIONS:
Overall Officials: Claude LAMBERT, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No